CLINICAL TRIAL: NCT02302833
Title: A Phase II Study to Evaluate the Effects of Cabozantinib in Patients With Unresectable Metastatic Pheochromocytomas and Paragangliomas
Brief Title: Cabozantinib S-malate in Treating Patients With Metastatic Pheochromocytomas or Paragangliomas That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0081; NCI-2014-02607 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0081 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-11-21; First posted 2014-11-27 (Estimated); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Paraganglioma; Metastatic Adrenal Gland Pheochromocytoma; Metastatic Paraganglioma; Regional Adrenal Gland Pheochromocytoma; Unresectable Adrenal Gland Pheochromocytoma; Unresectable Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabozantinib s-malate) (Experimental): Patients receive cabozantinib s-malate PO QD on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL-184; XL184
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot phase II trial studies how well cabozantinib s-malate works in treating patients with pheochromocytomas or paragangliomas that have spread from the primary site to other places in the body and cannot be removed by surgery. Cabozantinib s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking the growth of new blood vessels necessary for tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate best overall response rate in patients with measurable disease determined by computed tomography (CT) or magnetic resonance imaging (MRI).

SECONDARY OBJECTIVES:

I. To estimate progression-free survival at 1-year. II. To correlate blood pressure control and change/discontinuation of antihypertensive medications with tumor responses.

III. To correlate symptomatology evaluation by the MD Anderson Symptom Inventory (MDASI) with tumor responses.

IV. To correlate plasma metanephrines and chromogranin A with tumor responses. V. To correlate plasma C-reactive protein and interleukin-6 with symptoms and tumor responses.

VI. Toxicity assessment by the Common Terminology Criteria for Adverse Events (CTCAE).

VII. To correlate both c-MET expression by immunohistochemistry (IHC) as well as MET amplification by fluorescence in situ hybridization (FISH) in archived samples and correlate these biomarkers with overall prognosis and responsiveness to cabozantinib (cabozantinib s-malate).

EXPLORATORY OBJECTIVES:

I. Best overall response rate in patients with bone metastases only (8 patients) as determined by fludeoxyglucose F 18 positron emission tomography/computed tomography (FDG-PET/CT).

II. FDG-PET/CT maximum standard uptake value (SUVmax), advanced volumetric measures including peak standard uptake value (SUVpeak), metabolic tumor volume (MTV), and total lesion glycolysis (TLG).

III. Time to skeletal related events. IV. Incidence of skeletal related events at 4 months and one year. V. Markers of bone turnover (bone specific alkaline phosphatase and C-terminal telopeptide [CTx]).

OUTLINE:

Patients receive cabozantinib s-malate orally (PO) once daily (QD) on days 1-28. Courses repeat every 4 weeks through week 24 and then every 8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30-37 days.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of pheochromocytoma (PH)/paraganglioma (PG)
* Locally advanced or metastatic disease not amenable to surgery
* Patients enrolled in the main branch should have measurable disease; patients with a predominance of bone disease who have small, non-measurable or small measurable lesions other than bone, may be included per the principal investigator's discretion, in the exploratory branch of the study for patients with bone metastases only
* Progressive disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the investigator within the 12 months preceding study enrollment
* Assessment of all known disease sites, e.g., by CT scan, MRI, bone scan as appropriate, and/or FDG-PET scan within 28 days before the first dose of cabozantinib
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of at least 3 months
* Absolute neutrophil count (ANC) >= 1500/mm^3 without colony stimulating factor support (within 4 days prior to the first dose of cabozantinib)
* Platelets >= 100,000/mm^3 (within 4 days prior to the first dose of cabozantinib)
* Hemoglobin >= 9 g/dL (within 4 days prior to the first dose of cabozantinib)
* Bilirubin =< 1.5 x the upper limit of normal (ULN) (for subjects with known Gilbert's disease, bilirubin =< 3.0 mg/dL) (within 4 days prior to the first dose of cabozantinib)
* Serum albumin >= 2.8 g/dl (within 4 days prior to the first dose of cabozantinib)
* Serum creatinine =< 1.5 x ULN or creatinine clearance (CrCl) >= 50 mL/min (for creatinine clearance estimation, the Cockcroft and Gault equation should be used) (within 4 days prior to the first dose of cabozantinib)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 x ULN (within 4 days prior to the first dose of cabozantinib)
* Lipase < 2.0 x ULN and no radiologic or clinical evidence of pancreatitis (within 4 days prior to the first dose of cabozantinib)
* Urine protein/creatinine ratio (UPCR) =< 1 (within 4 days prior to the first dose of cabozantinib)
* Serum phosphorus, calcium, potassium >= lower limit of normal (LLN) (within 4 days prior to the first dose of cabozantinib)
* Serum magnesium >= 1.2 mg/dL (within 4 days prior to the first dose of cabozantinib)
* Capable of understanding and complying with the protocol requirements and has signed the informed consent document
* Sexually active patients (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used; all subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s)
* Women of childbearing potential must have a negative pregnancy test at screening; women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal; postmenopause is defined as amenorrhea >= 12 consecutive months; note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason

Exclusion Criteria:

* Received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 3 weeks, or nitrosoureas/mitomycin C within 6 weeks before the first dose of study treatment
* Prior treatment with cabozantinib
* Radiation therapy for bone metastasis within 2 weeks, or any other external radiation therapy within 4 weeks before the first dose of study treatment; subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Received radionuclide treatment (i.e. iodine [I]-131 meta-iodo-benzyl guanidine) within 6 months of the first dose of study treatment
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 14 days before the first dose of study treatment
* Receipt of any other type of investigational agent within 28 days before the first dose of study treatment
* The subject has not recovered to baseline or CTCAE =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs)
* Prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test >= 1.3 x the laboratory ULN within 7 days before the first dose of study treatment
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (eg, clopidogrel); low dose aspirin (=< 81 mg/day), low-dose warfarin (=< 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted
* The subject requires chronic concomitant treatment of strong cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's wort)
* The subject has experienced any of the following: a. clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment, b. hemoptysis of >= 0.5 teaspoon (2.5 ml) of red blood within 3 months before the first dose of study treatment, c. any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* Radiographic evidence of cavitating pulmonary lesion(s)
* Tumor invading or encasing any major blood vessels
* Evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* Uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions: a. cardiovascular disorders including: i. congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening, ii. concurrent uncontrolled hypertension defined as sustained blood pressure > 150 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment, iii. any history of congenital long QT syndrome, or iv. any of the following within 6 months before the first dose of study treatment: unstable angina pectoris, clinically-significant cardiac arrhythmias, stroke (including transient ischemic attack [TIA], or other ischemic event), myocardial infarction, or thromboembolic event requiring therapeutic anticoagulation (note: subjects with a venous filter [e.g. vena cava filter] are not eligible for this study)

  * Gastrointestinal disorders, particularly those associated with a high risk of perforation or fistula formation, including: i. any of the following within 28 days before the first dose of study treatment: intra-abdominal tumor/metastases invading GI mucosa, active peptic ulcer disease (patients must be completely recovered), inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis (patient must be completely recovered from these conditions), malabsorption syndrome; ii. any of the following within 6 months before the first dose of study treatment: abdominal fistula, gastrointestinal perforation, bowel obstruction or gastric outlet obstruction, or intra-abdominal abscess (complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment); c. other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy, d. other clinically significant disorders such as: i. active infection requiring systemic treatment within 28 days before the first dose of study treatment, ii. serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment, iii. history of organ transplant, iv. concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment, or v. major surgery within 12 weeks before the first dose of study treatment; complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment; minor surgery within 28 days before the first dose of study treatment with complete wound healing at least 10 days before the first dose of study treatment; subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Unable to swallow tablets
* A corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before first dose of study treatment; three electrocardiograms (ECGs) must be performed; if the average of these three consecutive results for QTcF is =< 500 msec, the subject meets eligibility in this regard
* Pregnant or breastfeeding
* A previously identified allergy or hypersensitivity to components of the study treatment formulation
* Unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* Evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment except for cured nonmelanoma skin cancer or cured in situ cervical carcinoma
* Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality which, in the judgment of the investigator, would have made the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Jimenez, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jimenez C, Habra MA, Campbell MT, Tamsen G, Cruz-Goldberg D, Long J, Bassett R, Dantzer R, Balderrama-Brondani V, Varghese J, Lu Y. Cabozantinib in patients with unresectable and progressive metastatic phaeochromocytoma or paraganglioma (the Natalie Trial): a single-arm, phase 2 trial. Lancet Oncol. 2024 May;25(5):658-667. doi: 10.1016/S1470-2045(24)00133-5. Epub 2024 Apr 9. PMID 38608693
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cabozantinib: Patients with advanced and progressive pheochromocytomas and paragangliomas meeting inclusion and exclusion criteria
  Patients receive cabozantinib s-malate PO QD on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
Period: Overall Study
Arm/Group | Cabozantinib
Started | 20
Completed | 17
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 52 [37 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 17
percentage of participants | 25 [7.3 to 52]

ADVERSE EVENTS:
Time Frame: 9 years
Arm/Group | Cabozantinib
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 20/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=20)
Abdominal pain (Gastrointestinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial infection (Infections and infestations) | 1
Chest Pain (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Gastrointestinal fistula (Gastrointestinal disorders) | 1
Heart Failure (Cardiac disorders) | 1
Heart Failure, Death (Cardiac disorders) | 1
Hypersomnia (General disorders) | 1
Hypertension (Vascular disorders) | 1
Left Ventricular systolic dysfunction (Cardiac disorders) | 1
Musculoskeletal and connective tissue disorder-other, Specify (Musculoskeletal and connective tissue disorders) | 1
Myelodysplastic Syndrome, Death (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral Hemorrhage (General disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Small Intestine obstruction (Gastrointestinal disorders) | 1
Stroke (Nervous system disorders) | 1
Surgical and medical Procedures Other, Laminectomy, Tumor resection (Surgical and medical procedures) | 1
Surgical and medical Procedures Other: Hip Replacement (Surgical and medical procedures) | 1
Surgical and medical Procedures Other: Laminectomy Sacrum (Surgical and medical procedures) | 1
Thromboembolic Event (Vascular disorders) | 2
Urinary Tract Infection (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=20)
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 8
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 7
Agitation (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 15
Alkaline phosphatase increased (Investigations) | 11
Allergic rhinitis (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 8
ALT increased (Investigations) | 1
Anal fistula (General disorders) | 1
Anal pain (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 18
Anorexia (Metabolism and nutrition disorders) | 13
Anxiety (Psychiatric disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 16
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9
Bloating (Gastrointestinal disorders) | 7
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 7
Blood bilirubin increased (Investigations) | 2
Blurred vision (Eye disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bruising (General disorders) | 5
Burn (Skin and subcutaneous tissue disorders) | 1
Buttock pain (General disorders) | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1
Chills (General disorders) | 1
Concentration impairment (Psychiatric disorders) | 4
Confusion (Psychiatric disorders) | 1
Conjunctivitis (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Cough (General disorders) | 7
Creatinine increased (Investigations) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 15
Dizziness (General disorders) | 8
Dry mouth (General disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 11
Dysgeusia (General disorders) | 13
Dyspepsia (General disorders) | 1
Dysphagia (General disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Ear and labyrinth disorders (Ear and labyrinth disorders) | 2
Edema limbs (General disorders) | 7
Electrocardiogram QT corrected interval prolonged (General disorders) | 2
Endocrine disorders (Endocrine disorders) | 3
Epistaxis (Vascular disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Extraocular muscle paresis (Musculoskeletal and connective tissue disorders) | 1
Eye disorders (Eye disorders) | 3
Eye pain (Eye disorders) | 2
Fall (General disorders) | 2
Fatigue (General disorders) | 19
Fecal incontinence (General disorders) | 1
Fever (General disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flatulence (Gastrointestinal disorders) | 3
Flu like symptoms (General disorders) | 4
Flushing (Vascular disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders (Gastrointestinal disorders) | 5
General disorders and administration site conditions (General disorders) | 13
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
GERD (Gastrointestinal disorders) | 1
Hand and foot syndrome (General disorders) | 1
Headache (Nervous system disorders) | 12
Heart Failure (Cardiac disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Hoarseness (General disorders) | 7
Hot flashes (General disorders) | 1
Hypercalcemia (Investigations) | 1
Hyperglycemia (Investigations) | 15
Hyperhidrosis (General disorders) | 11
Hyperkalemia (Investigations) | 2
Hypertension (Investigations) | 19
Hyperthyroidism (Investigations) | 1
Hyperuricemia (Investigations) | 1
Hypoalbuminemia (Investigations) | 7
Hypocalcemia (Investigations) | 3
Hypoglycemia (Investigations) | 2
Hypokalemia (Investigations) | 3
Hypomagnesemia (Investigations) | 8
Hyponatremia (Investigations) | 4
Hypophosphatemia (Investigations) | 4
Hypotension (General disorders) | 1
Hypothyroidism (Endocrine disorders) | 13
Immune system disorders (Immune system disorders) | 1
INR increased (Investigations) | 4
Insomnia (Psychiatric disorders) | 6
Investigations (Investigations) | 15
Irregular menstruation (Reproductive system and breast disorders) | 1
Irritability (General disorders) | 1
Laryngeal inflammation (Gastrointestinal disorders) | 1
LDH (General disorders) | 1
Libido decreased (General disorders) | 1
Lipase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 13
Memory impairment (Nervous system disorders) | 3
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1
Mucosal infection (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 13
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 1
Nail ridging (General disorders) | 1
Nasal congestion (General disorders) | 1
Nausea (Gastrointestinal disorders) | 15
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Nervous system disorders (Nervous system disorders) | 2
Neutrophil Abs Increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 1
Oral dysesthesia (Gastrointestinal disorders) | 2
Pain (General disorders) | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 13
Palpitations (Cardiac disorders) | 8
Paresthesia (General disorders) | 8
Paronychia (Skin and subcutaneous tissue disorders) | 2
Periorbital edema (Eye disorders) | 1
Pharyngeal mucositis (Gastrointestinal disorders) | 1
Photophobia (General disorders) | 1
Photosensitivity (General disorders) | 1
Platelet count decreased (Investigations) | 9
Platelet Count increased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Investigations) | 13
Psychiatric disorders (Psychiatric disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Rectal fistula (General disorders) | 1
Renal and urinary disorders (Renal and urinary disorders) | 2
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 6
Right hip cramp (Musculoskeletal and connective tissue disorders) | 1
Scalp pain (General disorders) | 1
Serum amylase increased (Investigations) | 3
Sinus Bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 5
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 15
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 5
Skin infection (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Somnolence (General disorders) | 1
Sore throat (General disorders) | 3
Stroke (Nervous system disorders) | 1
Surgical and medical procedures (Surgical and medical procedures) | 2
Thromboembolic event (Vascular disorders) | 2
Toothache (General disorders) | 5
U prot/Creat increased (Investigations) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 2
Urine color change (Renal and urinary disorders) | 1
Vasculitis (Vascular disorders) | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Watering eyes (Eye disorders) | 1
WBC count increased (Investigations) | 1
Weight loss (General disorders) | 17
White blood cell decreased (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT02302833/Prot_SAP_000.pdf